CLINICAL TRIAL: NCT02219087
Title: Local Liposomal Bupivacaine Versus Standard of Care in an Opioid-Sparing Analgesic Approach to Total Knee Arthroplasty: A Prospective, Randomized, Controlled Trial
Brief Title: Liposomal Bupivacaine Versus Standard of Care in Total Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, Robert Fada, MD, Orthopedic Surgeon, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0024
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee arthroplasty; Total joint arthroplasty; Knee replacement; Osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): Pre-operative adductor canal nerve block (20mL of 0.5% ropivacaine). Liposomal bupivacaine (diluted to 60mL): 20mL into the posterior pocket, 20mL into the lateral, and 20mL into the medial, including all deep and superficial tissues of these areas.
  Interventions: Drug: Liposomal bupivacaine
- Standard of Care (Active Comparator): Pre-operative adductor canal nerve block (20mL of 0.5% ropivacaine). Intra-operative popliteal nerve block from the surgeon: 20mL 0.2% ropivacaine and a peri-articular injection of 10mg morphine, 30mg ketorolac and 40mg methylprednisolone.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Standard of Care — Pre-operative adductor canal nerve block (20mL of 0.5% ropivacaine). Intra-operative popliteal nerve block from the surgeon: 20mL 0.2% ropivacaine and a peri-articular injection of 10mg morphine, 30mg ketorolac and 40mg methylprednisolone.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine whether liposomal bupivacaine is effective in the management of pain following total knee arthroplasty, as compared to standard of care analgesia.

DETAILED DESCRIPTION:
Liposomal bupivacaine (Exparel®) is a local anesthetic made up of liposomal encapsulated bupivacaine. It is designed to be injected at the time of surgery into the local soft tissues. Because of its unique liposomal delivery system, Liposomal bupivacaine (Exparel®) has been shown to provide up to 96 hours of pain relief following surgeries. This makes it an attractive option in total knee arthroplasty patients. Combined with the proven efficacy of regional anesthesia, intraoperative liposomal bupivacaine (Exparel®) may provide extended pain relief following total knee arthroplasty. This has the potential to avoid the need for opioid medications. With better pain control, medication side effects can be avoided and patient's length of stay in the hospital can be shortened.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Scheduled to undergo total knee arthroplasty (TKA) performed by the principal investigator

Exclusion Criteria:

* Age <18 years
* Pregnant or breastfeeding
* Non-English-speaking
* Unable to give informed consent
* Patients admitted from or discharged to a medical facility (due to likelihood of limited mobility and/or required minimum lengths of stay, confounding primary outcome), including other hospitals, skilled nursing facilities, long-term acute care hospitals, etc.
* Patients unable to complete a device-assisted 140 foot walk at baseline
* Patients with contraindication(s) to any bupivacaine or ropivacaine formulation, to nerve blocks or any of the local agents used (IV morphine, ketorolac, or methylprednisolone).
* Patients on a long-acting maintenance opioid prior to admission for surgery (e.g., methadone, oxycontin)
* Patients undergoing simultaneous bilateral TKAs, as this would increase the dose of Exparel per patient (we are limited to one dose per patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fada, MD, Principal Investigator — OhioHealth; Sara Jordan, PharmD, BCPS, Study Director — OhioHealth
Locations (1):
- OhioHealth Grant Medical Center Bone and Joint Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Pre-operative adductor canal nerve block (20mL of 0.5% ropivacaine). Liposomal bupivacaine (diluted to 60mL): 20mL into the posterior pocket, 20mL into the lateral, and 20mL into the medial, including all deep and superficial tissues of these areas.
  Liposomal bupivacaine
- Standard of Care: Pre-operative adductor canal nerve block (20mL of 0.5% ropivacaine). Intra-operative popliteal nerve block from the surgeon: 20mL 0.2% ropivacaine and a peri-articular injection of 10mg morphine, 30mg ketorolac and 40mg methylprednisolone.
  ropivacaine, morphine ,ketorolac, methylprednisolone: Standard of care analgesia
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Standard of Care
Started | 30 | 30
Completed | 30 | 29 (Randomization envelope pulled out of sequence for consented patient. Excluded by request of IRB)
Not Completed | 0 | 1
Not completed — Randomization envelope pulled out of seq | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Standard of Care | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (8.3) | 61.2 (8.9) | 63.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number Physical Therapy Sessions Necessary for Discharge
Description: Number of physical therapy (PT) sessions necessary for discharge. A significant decrease in the number of sessions will be defined as ≥ 2. Typically, there are 2 sessions per day, with each patient completing an average of 4-5 sessions during their admission.
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 2.5 days.
Measure: Mean (Standard Deviation); unit: Physical Therapy Sessions
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
Physical Therapy Sessions | 3.0 (1.2) | 3.6 (1.3)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard of Care; Test type: Superiority or Other; p = 0.137, t-test, 2 sided

2. Secondary Outcome: Mean Visual Analog Scale (VAS) Pain Scores During Hospital Stay
Description: VAS was measured using a scale that ranged from 0 to 10. Higher scores indicate more pain, or a worse outcome. Patients had pain measured a variable number of times following surgery before discharge. Mean VAS score during the hospital stay for each patient was calculated
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 2.5 days.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
Units on a scale | 4.4 (1.3) | 4.7 (1.5)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard of Care; Test type: Superiority or Other; p = 0.343, t-test, 2 sided

3. Secondary Outcome: Length of Stay (LOS, in Days)
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 2.5 days.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
Days | 2.5 (0.8) | 2.3 (0.5)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard of Care; Test type: Superiority or Other; p = 0.208, t-test, 2 sided

4. Secondary Outcome: Opioid Consumption in Oral Morphine Equivalents (OMEs, in Milligrams)
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 2.5 days.
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
Milligrams | 274.6 (121.0) | 304.8 (143.4)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard of Care; Test type: Superiority or Other; p = 0.385, t-test, 2 sided

5. Secondary Outcome: Number of Participants With Opioid-related Adverse Events (ORAEs) During Hospital Stay
Description: 1. Nausea
  2. Vomiting
  3. Constipation
  4. Ileus
  5. Pruritus
  6. Respiratory depression
  7. Over-sedation
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 2.5 days.
Measure: Number; unit: participants
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
participants | 13 | 11
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard of Care; Test type: Superiority or Other; p = 0.843, Chi-squared

6. Secondary Outcome: Total Cost of Care (Dollars)
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 2.5 days.
Measure: Median (Full Range); unit: Dollars
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
Dollars | 64582.90 [55424.50 to 121583.50] | 62601.50 [52435.90 to 97367.50]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Standard of Care; Test type: Superiority or Other; p = 0.438, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Hospital Readmission Not Including Admissions Planned Procedures
Time Frame: Participants will be followed for 30 days after leaving the hospital.
Measure: Number; unit: participants
Arm/Group | Liposomal Bupivacaine | Standard of Care
Number analyzed (Participants) | 30 | 29
participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 13/30 | 11/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine (N=30) | Standard of Care (N=29)
Nausea/Vomiting (Gastrointestinal disorders) | 10 | 9
Constipation (Gastrointestinal disorders) | 6 | 4
Oversedation (Nervous system disorders) | 4 | 0
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes